CLINICAL TRIAL: NCT01641367
Title: Management Using the Latest Technologies in Resource-limited Settings to Optimize Combination Therapy After Viral Failure (MULTI-OCTAVE)
Brief Title: A5288/MULTI-OCTAVE: Management Using Latest Technologies to Optimize Combination Therapy After Viral Failure
Acronym: MULTI-OCTAVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); AbbVie (Industry); Gilead Sciences (Industry); Janssen Pharmaceuticals (Industry); Merck Sharp & Dohme LLC (Industry); Dimagi Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5288; 1U01AI068636 (NIH)
Record Dates: First submitted 2012-06-28; First posted 2012-07-16 (Estimated); Results first posted 2018-02-20 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Darunavir; etravirine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Raltegravir Potassium; bactericidal permeability increasing protein; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort A (Experimental): Under Protocol version 1.0:
  No resistance to NRTIs, PIs, or NNRTI
  • Continue current second-line regimen; NRTIs could be modified
  Changed under LOA#2 to:
  No LPV/RTV resistance and susceptible to at least one NRTI, regardless of NNRTI resistance or prior RAL exposure
  • Continue second-line regimen which may include LPV/RTV; NRTIs could be modified
  Changed under LOA#3 to:
  No LPV/RTV resistance and susceptible to at least one NRTI, regardless of NNRTI resistance or prior RAL exposure
  • Continue PI backbone; NRTIs could be modified. If on a RAL-containing regimen, RAL must be discontinued.
  Interventions: Drug: Second line ART regimens - based on a boosted protease inhibitor (bPI) plus two nucleoside analogues (NRTIs); Other: SOC adherence versus SOC+CPI adherence
- Sub-cohort B1 (Experimental): Under Protocol version 1.0:
  Susceptible to DRV/RTV and ETR with or without resistance to NRTIs (and may have resistance to other PIs) and without active hepatitis B infection at screening
  • Best available NRTIs, RAL, & DRV/RTV
  Changed under LOA#2 to:
  Resistance to LPV/RTV but susceptible to DRV/RTV and ETR and with no prior RAL exposure and regardless of NRTI resistance (and without active hepatitis B infection at screening) OR Resistance to all NRTIs (i.e. susceptible to none) but susceptible to DRV/RTV and ETR and with no prior RAL exposure (and without active hepatitis B infection at screening)
  • Best available NRTIs, RAL, & DRV/RTV
  Interventions: Drug: Darunavir; Drug: Raltegravir; Other: SOC adherence versus SOC+CPI adherence
- Sub-cohort B2 (Experimental): Under Protocol version 1.0:
  Susceptible to DRV/RTV and ETR with or without resistance to NRTIs (and may have resistance to other PIs) and without active hepatitis B infection at screening
  • ETR, RAL, and DRV/RTV
  Changed under LOA#2 to:
  Resistance to LPV/RTV but susceptible to DRV/RTV and ETR and with no prior RAL exposure and regardless of NRTI resistance (and without active hepatitis B infection at screening) OR Resistance to all NRTIs (i.e. susceptible to none) but susceptible to DRV/RTV and ETR and with no prior RAL exposure (and without active hepatitis B infection at screening)
  • ETR, RAL, and DRV/RTV
  Interventions: Drug: Darunavir; Drug: Etravirine; Drug: Raltegravir; Other: SOC adherence versus SOC+CPI adherence
- Sub-cohort B3 (Experimental): Under Protocol version 1.0:
  Susceptible to DRV/RTV and ETR with or without resistance to NRTIs (and may have resistance to other PIs) and with active hepatitis B infection at screening
  • RAL, DRV/RTV, and FTC/TDF or TDF+3TC
  Changed under LOA#2 to:
  Resistance to LPV/RTV but susceptible to DRV/RTV and ETR and with no prior RAL exposure and regardless of NRTI resistance (with active hepatitis B infection at screening) OR Resistance to all NRTIs (i.e. susceptible to none) but susceptible to DRV/RTV and ETR and with no prior RAL exposure (with active hepatitis B infection at screening)
  • RAL, DRV/RTV, and FTC/TDF or TDF+3TC
  Interventions: Drug: Darunavir; Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Raltegravir; Other: SOC adherence versus SOC+CPI adherence
- Cohort C (Experimental): Under Protocol version 1.0:
  Resistance to NRTIs and ETR or resistance to ETR alone (and may have resistance to PIs other than DRV)
  • Best available NRTIs, RAL, and DRV/RTV
  Changed under LOA#2:
  Resistance to LPV/RTV and ETR but susceptible to DRV/RTV and with no prior RAL exposure and regardless of NRTI resistance OR Resistance to ETR and to all NRTIs (i.e. susceptible to none) but susceptible to DRV/RTV and with no prior RAL exposure
  • Best available NRTIs, RAL, and DRV/RTV
  Interventions: Drug: Darunavir; Drug: Raltegravir; Other: SOC adherence versus SOC+CPI adherence
- Cohort D (Experimental): Under Protocol version 1.0:
  Multiple NRTI resistance and/or DRV/RTV resistance or prior RAL exposure:
  • Best available regimen, including study-provided and any locally available drugs
  Changed under LOA#2:
  Not eligible for Cohort A, B, or C:
  • Best available regimen, including study-provided and any locally available drugs
  Updated under protocol v2.0:
  • Best available ART regimen, including study-provided and any locally available non-experimental drugs
  Interventions: Drug: Study provided drugs according to patient resistance profile (DRV, ETR, RTV, FTC/TDF) + any in country available drug as applicable & available; Other: SOC adherence versus SOC+CPI adherence

INTERVENTIONS:
Drug: Darunavir — Participants were administered darunavir orally as one 600 mg tablet twice a day (1200 mg per day) with food (taken with Ritonavir 100 mg twice a day [200 mg per day])
  Other Names: DRV; Prezista
  Arms: Cohort C; Sub-cohort B1; Sub-cohort B2; Sub-cohort B3
Drug: Etravirine — Patients were administered Etravirine orally as two 100 mg tablets or one 200 mg tablet twice a day (400 mg per day) following a meal.
  Other Names: ETR; Intelence
  Arms: Sub-cohort B2
Drug: Emtricitabine/tenofovir disoproxil fumarate — Patients were administered FTC/TDF orally as one fixed dose combination tablet (FTC 200 mg/TDF 300 mg) once daily, with or without food.
  Other Names: FTC/TDF; Truvada
  Arms: Sub-cohort B3
Drug: Raltegravir — Participants were administered Raltegravir orally as one 400 mg tablet twice daily (800 mg per day), with or without food
  Other Names: RAL; Isentress
  Arms: Cohort C; Sub-cohort B1; Sub-cohort B2; Sub-cohort B3
Drug: Second line ART regimens - based on a boosted protease inhibitor (bPI) plus two nucleoside analogues (NRTIs) — LPV/r and ATV/r were the preferred bPIs for second-line ART. TDF + (3TC or FTC) or AZT + 3TC were the most frequent NRTI backbones. Cohort A did not include any of the new drugs; therefore, it is distinct from Cohorts B, C, and D.
  Arms: Cohort A
Drug: Study provided drugs according to patient resistance profile (DRV, ETR, RTV, FTC/TDF) + any in country available drug as applicable & available — For Cohort D, in many situations a participant received the same regimen that patients are getting in Cohorts B and C if that was the best combination that can be obtained according to his/her resistance profile and drug availability (as for many countries there were no further drug options beyond the available study drugs).
  Arms: Cohort D
Other: SOC adherence versus SOC+CPI adherence — * not participating in the adherence randomization; OR
  * randomized to SOC adherence; OR
  * randomized to SOC+CPI adherence.

SUMMARY:
The study was done to:

* test a strategy of using a resistance test to choose anti-HIV drugs
* see how well combinations of new anti-HIV drugs work to lower HIV infection
* see if taking new anti-HIV drugs together is safe and tolerable
* see if text messages improve people's anti-HIV drug-taking behavior (only at sites participating in the adherence study)
* in people taking certain combinations of anti-HIV drugs with an anti-TB drug, compare how these drugs act in the body
* to see how people do after they stop having frequent clinic visits as part of a research study

DETAILED DESCRIPTION:
A5288 was an open-label phase IV, prospective interventional, strategy study in resource-limited settings (RLS) for HIV-1 infected participants with triple-class experience or resistance to nucleoside reverse transcriptase inhibitors (NRTIs), non-NRTIs (NNRTIs), and protease inhibitors (PIs) and who were failing their current regimen. The use of novel agents and contemporary clinical decision management tools that include standard genotyping and plasma HIV viral load (VL) monitoring were evaluated. The screening genotype results and antiretroviral (ARV) history were used to allocate potential participants to one of four Cohorts (A, B, C or D) and to select an associated ARV regimen based on the Cohort assignment. In brief, individuals assigned to Cohort A continued on the same PI as in their second-line regimen, with the ability to modify NRTIs. Those assigned to Cohort B who were negative for hepatitis B were randomized to receive RAL and DRV/RTV with either the best available NRTIs (Cohort B1) or ETR (Cohort B2). If they were positive for hepatitis B they were assigned to Cohort B3 and received RAL, DRV/RTV and either FTC/TDF or 3TC/TDF. Individuals assigned to Cohort C received RAL and DRV/RTV with the best available NRTIs. Those ineligible for Cohorts A, B or C were assigned to Cohort D and received the best available regimen that included study provided drugs and any locally provided drugs.

At sites where feasible and relevant, the study evaluated an adherence support intervention. This involved a randomized comparison of a cell phone-based adherence support intervention plus local standard-of-care adherence support procedures (CPI+SOC) versus the SOC adherence support procedures.

Participants enrolled to the study in Step 1. If a participant experienced a confirmed virologic failure (defined as two consecutive HIV-1 RNA measures >= 1000 copies/mL) at/after 22 weeks on their Step 1 regimen, they had another genotype test performed and cohort/regimen selected for Step 2. With the exception of one additional visit 4 weeks after enrollment to Step 2, the visit schedule for Step 2 followed the participant's original Step 1 schedule throughout the remainder of follow up.

Participants were followed in Steps 1 and 2 until 48 weeks after the last participant was enrolled to Step 1. During the first 48 weeks after Step 1 enrollment, clinic visits occurred at weeks 4, 12, 24, 36 and 48. After week 48, visits occurred every 12 weeks for adherence, safety and efficacy measures.

Participants had a final step 1/2 visit between November 22, 2016 and February 13, 2017. At the final step 1/2 visit, participants taking RAL, ETR, or DRV who were unable to obtain these drugs locally (e.g., through local treatment programs), and were otherwise eligible, entered Step 3 and continued to receive these drugs through the study for up to 96 additional weeks. Step 3 participants were dispensed ARVs every 12 weeks and had clinical assessments every 24 weeks. The purpose of Step 3 was to assist participants with the transition back to local care.

The primary analysis specified in the protocol and in the Statistical Analysis Plan was to estimate the proportion of participants in the overall study population who were virologically suppressed (HIV-1 RNA ≤200 copies/mL) at week 48 with a 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria for Step 1:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA VL.
* Any previous combination of ARV treatment at any time with at least one regimen that contained one NNRTI and two NRTIs which was replaced with a PI-based regimen because of virologic, immunologic, or clinical treatment failure, or because of toxicity.

NOTE: All potential participants with prior RAL exposure were assigned to either Cohort A or Cohort D.

* At screening, receipt of a PI-based regimen with no regimen change for a minimum of 24 weeks prior to screening.
* Confirmation of VF of current second-line PI-based ART. NOTE A: Failure of the current second-line regimen was defined as two consecutive measurements of plasma HIV-1 RNA ≥1000 copies/mL obtained at least 1 day apart while on the current PI-based regimen. "Current PI-based regimen" and "current regimen" were understood to be the regimen described (ie, the regimen that the candidate was taking when the first VF sample was drawn plus only those modifications allowed).
* CD4+ T-cell count result from a specimen drawn within 103 days prior to study entry
* Laboratory values obtained within 30 days prior to study entry:

  * Absolute neutrophil count (ANC) ≥ 500/mm^3
  * Hemoglobin ≥7.5 g/dL
  * Platelet count ≥40,000/mm^3
  * Creatinine ≤2 X upper limit of normal (ULN)
  * Aspartate aminotransferase (AST), serum glutamic oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT), serum glutamic pyruvic transaminase (SGPT), and alkaline phosphatase ≤5 x ULN
  * Total bilirubin ≤2.5 x ULN
  * Creatinine clearance (CrCl) >30 mL/min, either measured or estimated by Cockcroft-Gault equation
  * Hepatitis B panel that includes HbsAB, HBcAB, and HBsAG or only HBsAG, with plasma stored for later anti-HBs and anti-HBc.

NOTE A: Candidates who were eligible for cohort B and who were positive for active hepatitis B infection were assigned to sub-cohort B3 at registration/randomization.

NOTE B: Candidates with CrCl <60 mL/min who were also positive for active hepatitis B infection were not eligible.

* Females of reproductive potential (women who have not been post-menopausal for at least 24 consecutive months, ie, who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, hysterectomy or bilateral salpingectomy or bilateral oophorectomy or tubal ligation) must have had a negative serum or urine pregnancy test prior to the submission of the screening genotype testing sample and again within 48 hours prior to randomization or registration.
* Female participants of reproductive potential must have agreed not to participate in the conception process (ie, active attempt to become pregnant, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the female participant must have used at least one reliable form of contraceptive. Female participants must have continued to use contraceptives while receiving study treatment and for 6 weeks after stopping study treatment.

Acceptable forms of contraceptives included:

* Condoms (male or female) with or without a spermicidal agent
* Diaphragm or cervical cap with spermicide
* Intrauterine device (IUD)
* Hormonal contraception

Female participants who were not of reproductive potential or whose male partner(s) had documented azoospermia) were not required to use contraceptives. Any statement of self-reported sterility or that of her partner's must have been entered in the source documents.

NOTE: Acceptable documentation of lack of reproductive potential was oral or written documentation from the participant.

* Karnofsky performance score >/= 70 within 30 days prior to study entry.
* Ability and willingness of potential participant to provide informed consent.
* Willingness of potential participant to adhere to protocol requirements, especially with respect to treatment assignment and ability to obtain non-study provided ART, if needed.
* Ability to take oral study medications.
* No intention of permanent relocation that would preclude attending Step 1 and 2 study follow-up visits.
* Availability of a successful, interpretable resistance genotype report from a DAIDS-approved regional genotyping facility from testing performed on a plasma sample that was collected during screening (ie, at or after the date that a sample is collected to confirm HIV-1 virologic failure) and which was shipped to a regional resistance testing laboratory once documentation of two screening plasma HIV-1 RNA values ≥1000 copies/mL were available.
* Identification of a cohort assignment and ARV regimen for use on study, selected from the recommended options provided by the site investigator, and reviewed and approved by the A5288 Clinical Management Committee (CMC).

Exclusion Criteria for Step 1:

* Pregnancy or breast-feeding.
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would have interfered with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization until candidate either completes therapy or was clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry.
* Concurrent illness or condition that would compromise the ability to take study medication, follow the protocol, or that would make participation not in the best interest of the participant, per the site investigator.
* Requirement for taking any of the prohibited medications with the selected ARV study regimen, or within 14 days prior to study entry.

NOTE: Study candidates should not have discontinued any component of their ART during screening. The 14-day restriction on prohibited medications did not apply to ARVs.

* Active tuberculosis (TB) or rifampin exposure less than 2 weeks prior to study entry.
* Any exposure to darunavir or etravirine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Grinsztejn, MD, PhD, Study Chair — Instituto de Pesquisa Clinica Evandro Chagas-Fiocruz; Peter Mugyenyi, MB ChB, FRCP, DSc, Study Chair — Joint Clinical Research Center
Locations (19):
- Brazil (2):
  - Hospital Nossa Senhora da Conceicao CRS (12201), Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro
- Haiti (2):
  - Les Centres GHESKIO CRS (30022), Port-au-Prince, Bicentaire
  - GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS, Port-au-Prince
- India (2):
  - BJ Medical College CRS (31441), Pune, Maharashtra
  - Chennai Antiviral Research and Treatment (CART) CRS (11701), Chennai, Taramani
- Kenya (2):
  - AMPATH at Moi Univ. Teaching Hosp. Eldoret CRS (12601), Eldoret
  - Kenya Medical Research Institute/Center for Disease Control (KEMRI/CDC) CRS (31460), Kisumu
- Malawi CRS (12001), Lilongwe, Malawi
- Peru (2):
  - San Miguel CRS (11302), San Miguel, Lima region
  - Barranco CRS (11301), Lima
- South Africa (4):
  - University of the Witwatersrand Helen Joseph (WITS HJH) CRS (11101), Johannesburg, Gauteng
  - Family Clinical Research Unit (FAM-CUR) CRS (8950), Cape Town, West Cape
  - Durban Adult HIV CRS (11201), Durban
  - Soweto ACTG CRS (12301), Johannesburg
- Thailand (2):
  - 31802 Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Bangkok, Patumwan
  - 31784 Chiang Mai University HIV Treatment CRS, Chiang Mai
- JCRC CRS, Kampala, Uganda
- UZ-Parirenyatwa CRS (30313), Harare, Zimbabwe

REFERENCES:
- [Derived] Avihingsanon A, Hughes MD, Salata R, Godfrey C, McCarthy C, Mugyenyi P, Hogg E, Gross R, Cardoso SW, Bukuru A, Makanga M, Badal-Aesen S, Mave V, Ndege BW, Fontain SN, Samaneka W, Secours R, Van Schalkwyk M, Mngqibisa R, Mohapi L, Valencia J, Sugandhavesa P, Montalban E, Munyanga C, Chagomerana M, Santos BR, Kumarasamy N, Kanyama C, Schooley RT, Mellors JW, Wallis CL, Collier AC, Grinsztejn B; A5288 Study team. Third-line antiretroviral therapy, including raltegravir (RAL), darunavir (DRV/r) and/or etravirine (ETR), is well tolerated and achieves durable virologic suppression over 144 weeks in resource-limited settings: ACTG A5288 strategy trial. J Int AIDS Soc. 2022 Jun;25(6):e25905. doi: 10.1002/jia2.25905. PMID 36039892
- [Derived] Godfrey C, Hughes MD, Ritz J, Coelho L, Gross R, Salata R, Mngqibisa R, Wallis CL, Mumbi ME, Matoga M, Poongulali S, Van Schalkwyk M, Hogg E, Fletcher CV, Grinsztejn B, Collier AC; A5288 team. Brief Report: Sex Differences in Outcomes for Individuals Presenting for Third-Line Antiretroviral Therapy. J Acquir Immune Defic Syndr. 2020 Jun 1;84(2):203-207. doi: 10.1097/QAI.0000000000002324. PMID 32049773
- [Derived] Gross R, Ritz J, Hughes MD, Salata R, Mugyenyi P, Hogg E, Wieclaw L, Godfrey C, Wallis CL, Mellors JW, Mudhune VO, Badal-Faesen S, Grinsztejn B, Collier AC. Two-way mobile phone intervention compared with standard-of-care adherence support after second-line antiretroviral therapy failure: a multinational, randomised controlled trial. Lancet Digit Health. 2019 May;1(1):e26-e34. doi: 10.1016/S2589-7500(19)30006-8. Epub 2019 May 6. PMID 31528850
- [Derived] Grinsztejn B, Hughes MD, Ritz J, Salata R, Mugyenyi P, Hogg E, Wieclaw L, Gross R, Godfrey C, Cardoso SW, Bukuru A, Makanga M, Faesen S, Mave V, Wangari Ndege B, Nerette Fontain S, Samaneka W, Secours R, van Schalkwyk M, Mngqibisa R, Mohapi L, Valencia J, Sugandhavesa P, Montalban E, Avihingsanon A, Santos BR, Kumarasamy N, Kanyama C, Schooley RT, Mellors JW, Wallis CL, Collier AC; A5288 Team. Third-line antiretroviral therapy in low-income and middle-income countries (ACTG A5288): a prospective strategy study. Lancet HIV. 2019 Sep;6(9):e588-e600. doi: 10.1016/S2352-3018(19)30146-8. Epub 2019 Jul 29. PMID 31371262
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004; Clarification, August 2009 — https://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf?sfvrsn=6
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=10

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between 22FEB2013 and 21DEC2015 at non-US based clinical research sites.
Groups:
- Experimental: Cohort A: Under Protocol version 1.0:
  No resistance to NRTIs, PIs, or NNRTI
  • Continue current second-line regimen; NRTIs could be modified
  Changed under LOA#2 to:
  No LPV/RTV resistance and susceptible to at least one NRTI, regardless of NNRTI resistance or prior RAL exposure • Continue second-line regimen which may include LPV/RTV; NRTIs could be modified
  Changed under LOA#3 to:
  No LPV/RTV resistance and susceptible to at least one NRTI, regardless of NNRTI resistance or prior RAL exposure
  • Continue PI backbone; NRTIs could be modified. If on a RAL-containing regimen, RAL must be discontinued.
- Experimental: Sub-cohort B1: Under Protocol version 1.0:
  Susceptible to DRV/RTV and ETR with or without resistance to NRTIs (and may have resistance to other PIs) and without active hepatitis B infection at screening • Best available NRTIs, RAL, & DRV/RTV
  Changed under LOA#2 to:
  Resistance to LPV/RTV but susceptible to DRV/RTV and ETR and with no prior RAL exposure and regardless of NRTI resistance (and without active hepatitis B infection at screening) OR Resistance to all NRTIs (i.e. susceptible to none) but susceptible to DRV/RTV and ETR and with no prior RAL exposure (and without active hepatitis B infection at screening)
  • Best available NRTIs, RAL, & DRV/RTV
- Experimental: Sub-cohort B2: Under Protocol version 1.0:
  Susceptible to DRV/RTV and ETR with or without resistance to NRTIs (and may have resistance to other PIs) and without active hepatitis B infection at screening • ETR, RAL, and DRV/RTV
  Changed under LOA#2 to:
  Resistance to LPV/RTV but susceptible to DRV/RTV and ETR and with no prior RAL exposure and regardless of NRTI resistance (and without active hepatitis B infection at screening) OR Resistance to all NRTIs (i.e. susceptible to none) but susceptible to DRV/RTV and ETR and with no prior RAL exposure (and without active hepatitis B infection at screening)
  • ETR, RAL, and DRV/RTV
- Experimental: Sub-cohort B3: Under Protocol version 1.0:
  Susceptible to DRV/RTV and ETR with or without resistance to NRTIs (and may have resistance to other PIs) and with active hepatitis B infection at screening • RAL, DRV/RTV, and FTC/TDF or TDF+3TC
  Changed under LOA#2 to:
  Resistance to LPV/RTV but susceptible to DRV/RTV and ETR and with no prior RAL exposure and regardless of NRTI resistance (with active hepatitis B infection at screening) OR Resistance to all NRTIs (i.e. susceptible to none) but susceptible to DRV/RTV and ETR and with no prior RAL exposure (with active hepatitis B infection at screening)
  • RAL, DRV/RTV, and FTC/TDF or TDF+3TC
- Experimental: Cohort C: Under Protocol version 1.0:
  Resistance to NRTIs and ETR or resistance to ETR alone (and may have resistance to PIs other than DRV) • Best available NRTIs, RAL, and DRV/RTV
  Changed under LOA#2:
  Resistance to LPV/RTV and ETR but susceptible to DRV/RTV and with no prior RAL exposure and regardless of NRTI resistance OR Resistance to ETR and to all NRTIs (i.e. susceptible to none) but susceptible to DRV/RTV and with no prior RAL exposure
  • Best available NRTIs, RAL, and DRV/RTV
- Experimental: Cohort D: Under Protocol version 1.0:
  Multiple NRTI resistance and/or DRV/RTV resistance or prior RAL exposure:
  • Best available regimen, including study-provided and any locally available drugs
  Changed under LOA#2:
  Not eligible for Cohort A, B, or C:
  • Best available regimen, including study-provided and any locally available drugs
  Updated under protocol v2.0:
  • Best available ART regimen, including study-provided and any locally available non-experimental drugs
- Cell Phone Intervention (CPI) + Standard of Care (SOC): The CPI was a simple interactive system (Short Message Service [SMS] Reminder and Flashback System) to identify non-adherence soon after it occurred and, in response, a site-based culturally relevant algorithm for managing barriers to adherence. Reminders were sent daily for the first 8 weeks on study, then three times per week for the next 8 weeks, and then weekly through to 48 weeks after study entry. Participants were expected to respond ("flashback") to each reminder. Failure to respond, triggered the system to alert the site to contact the participant. Sites were instructed to contact the participant if they missed any three flashbacks over two weeks during the daily messaging period, any two missed flashbacks over two weeks of the three times a week messaging period, and any two missed flashbacks over two weeks during the weekly messaging period. Additionally, sites were instructed to continue the local standard of care practices for managing adherence barriers.
- Standard of Care (SOC): Sites were instructed to continue the local standard of care practices for managing adherence barriers.
Period: Cohorts
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Started (Participants were followed on step 1/2 until 48 weeks after the last participant enrolled to Step 1.) | 287 | 74 | 72 | 8 | 70 | 34 | 0 | 0
Followed 72 Weeks on Step 1/2 | 211 | 60 | 60 | 6 | 52 | 30 | 0 | 0
Completed (Completed the study = participant must have had the last step 1/2 visit between 22NOV2016-13FEB2017) | 253 | 73 | 68 | 8 | 67 | 33 | 0 | 0
Not Completed | 34 | 1 | 4 | 0 | 3 | 1 | 0 | 0
Not completed — Death | 18 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 16 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Period: Randomized Adherence Intervention
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Started (Participants were followed on step 1/2 until 48 weeks after the last participant enrolled to Step 1.) | 0 | 0 | 0 | 0 | 0 | 0 | 257 | 264
Followed 72 Weeks on Step 1/2 | 0 | 0 | 0 | 0 | 0 | 0 | 196 | 202
Completed (Completed the study = participant must have had the last step 1/2 visit between 22NOV2016-13FEB2017) | 0 | 0 | 0 | 0 | 0 | 0 | 238 | 240
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 24
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 12
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 12

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D | Total
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34 | 545
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11) | 42 (10) | 42 (9) | 40 (10) | 42 (10) | 42 (10) | 41 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 29 | 28 | 4 | 23 | 14 | 258
  Male | 127 | 45 | 44 | 4 | 47 | 20 | 287
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 7 | 9 | 0 | 1 | 8 | 63
  Not Hispanic or Latino | 241 | 62 | 59 | 8 | 60 | 24 | 454
  Unknown or Not Reported | 8 | 5 | 4 | 0 | 9 | 2 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 62 | 21 | 17 | 3 | 35 | 8 | 146
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 195 | 49 | 49 | 5 | 34 | 21 | 353
  White | 7 | 1 | 3 | 0 | 0 | 3 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 23 | 3 | 3 | 0 | 1 | 1 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 25 | 8 | 8 | 0 | 0 | 8 | 49
  Haiti | 34 | 3 | 5 | 1 | 2 | 0 | 45
  India | 55 | 18 | 16 | 2 | 32 | 5 | 128
  Kenya | 32 | 9 | 8 | 1 | 7 | 2 | 59
  Malawi | 18 | 6 | 2 | 0 | 9 | 2 | 37
  Peru | 18 | 2 | 1 | 0 | 1 | 0 | 22
  South Africa | 58 | 7 | 11 | 0 | 7 | 1 | 84
  Thailand | 7 | 3 | 1 | 1 | 3 | 3 | 18
  Uganda | 34 | 13 | 17 | 2 | 6 | 9 | 81
  Zimbabwe | 6 | 5 | 3 | 1 | 3 | 4 | 22
Plasma HIV-1 RNA, categorical [Count of Participants; unit: Participants] — Baseline Plasma HIV-1 RNA is defined as the last available result on or before the date of study entry
  Participants
    < 40 copies/mL | 11 | 1 | 0 | 0 | 0 | 0 | 12
    40 - < 200 copies/mL | 11 | 2 | 1 | 1 | 2 | 1 | 18
    200 - < 1000 copies/mL | 32 | 5 | 3 | 1 | 9 | 2 | 52
    1000 - < 10,000 copies/mL | 59 | 17 | 20 | 3 | 12 | 10 | 121
    10,000 - < 100,000 copies/mL | 106 | 21 | 18 | 1 | 20 | 9 | 175
    100,000 - < 1,000,000 copies/mL | 60 | 27 | 25 | 2 | 22 | 10 | 146
    1,000,000 - < 10,000,000 copies/mL | 8 | 1 | 4 | 0 | 5 | 2 | 20
    >= 10,000,000 copies/mL | 0 | 0 | 1 | 0 | 0 | 0 | 1
CD4+ T-Cell Count, categorical [Count of Participants; unit: Participants] — Baseline CD4+ T-cell count is defined as the last available result on or before the date of study entry
  Participants
    < 50 cells/mm^3 | 50 | 17 | 11 | 1 | 9 | 7 | 95
    50 - < 200 cells/mm^3 | 108 | 27 | 25 | 1 | 31 | 10 | 202
    200 - < 350 cells/mm^3 | 79 | 15 | 23 | 5 | 19 | 7 | 148
    350 - < 500 cells/mm^3 | 30 | 12 | 6 | 1 | 6 | 8 | 63
    >= 500 cells/mm^3 | 20 | 3 | 7 | 0 | 5 | 2 | 37
IV drug history, categorical [Count of Participants; unit: Participants]
  Never | 286 | 74 | 72 | 8 | 70 | 34 | 544
  Previously | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis B Surface Antigen Result, categorical [Count of Participants; unit: Participants]
  Positive | 14 | 0 | 0 | 8 | 3 | 4 | 29
  Negative | 273 | 74 | 72 | 0 | 66 | 30 | 515
  Indeterminate | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Plasma HIV-1 RNA ≤200 Copies/mL at 48 Weeks
Description: The measurement closest to exactly 48 weeks (ie, 7x48=336 days) after the date of entry, within the window of 48 weeks ± 6 weeks (specifically 295 to 378 days after randomization, inclusive).
  The analysis in the protocol and in the Stat. Analysis Plan involved estimating the proportion of participants in the overall study population with HIV-1 RNA ≤200 copies/mL at week 48 with a 95% confidence interval calculated via a Wald approach. Death or lost to follow-up before week 48 was considered as HIV-1 RNA>200 copies/mL at week 48. Missing results at week 48 were considered as HIV-1 RNA >200 copies/mL at week 48 unless the immediately preceding and succeeding HIV-1 RNA measurements were ≤200 copies/mL. Since the primary analysis was on the total study population, overall results were also submitted. All participants in B3 had HIV-1 RNA ≤200 copies/mL at week 48. Therefore, Wald confidence interval could not be computed for B3 and Clopper-Pearson Exact confidence interval is provided.
Time Frame: 48 weeks after the date of entry
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Overall Study: Entire enrolled population spanning all arms and interventions.
Arm/Group | Overall Study | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 545 | 287 | 74 | 72 | 8 | 70 | 34
proportion of participants | 0.64 [0.60 to 0.68] | 0.44 [0.38 to 0.49] | 0.88 [0.80 to 0.95] | 0.88 [0.80 to 0.95] | 1.00 [0.63 to 1.00] | 0.90 [0.83 to 0.97] | 0.74 [0.59 to 0.88]

2. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA ≤200 Copies/mL at 24 Weeks
Description: The measurement closest to exactly 24 weeks (ie, 7x24=168 days) after the date of entry, within the window of 24 weeks ± 6 weeks (specifically 127 to 210 days after randomization, inclusive).
  The analysis in the protocol and in the Stat. Analysis Plan involved estimating the proportion of participants in the overall study population with HIV-1 RNA ≤200 copies/mL at week 24 with a 95% confidence interval calculated via a Wald approach. Death or lost to follow-up before week 24 was considered as HIV-1 RNA>200 copies/mL at week 24. Missing results at week 24 were considered as HIV-1 RNA >200 copies/mL at week 24 unless the immediately preceding and succeeding HIV-1 RNA measurements were ≤200 copies/mL. Since the primary analysis was on the total study population, overall results were also submitted. All participants in B3 had HIV-1 RNA ≤200 copies/mL at week 24. Therefore, Wald confidence interval could not be computed for B3 and Clopper-Pearson Exact confidence interval is provided.
Time Frame: 24 weeks after the date of entry
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Overall Study | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 545 | 287 | 74 | 72 | 8 | 70 | 34
proportion of participants | 0.64 [0.60 to 0.68] | 0.43 [0.37 to 0.48] | 0.89 [0.82 to 0.96] | 0.88 [0.80 to 0.95] | 1.00 [0.63 to 1.00] | 0.90 [0.83 to 0.97] | 0.74 [0.59 to 0.88]

3. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA ≤200 Copies/mL at 72 Weeks
Description: The measurement closest to exactly 72 weeks (ie, 7x72=504 days) after the date of entry, within the window of 72 weeks ± 6 weeks (specifically 463 to 546 days, inclusive).
  The analysis in the protocol and in the Analysis Plan involved estimating the proportion of participants in the overall study population with HIV-1 RNA ≤200 copies/mL at week 72 with a 95% confidence interval calculated via a Wald approach. Death or lost to follow-up before week 72 was considered as HIV-1 RNA>200 copies/mL at week 72. If a result was expected, missing results at week 72 were considered as HIV-1 RNA >200 copies/mL at week 72 unless the immediately preceding and succeeding HIV-1 RNA measurements were ≤200 copies/mL. Since the primary analysis was on the total study population, overall results were also submitted. All participants in B3 had HIV-1 RNA ≤200 copies/mL at week 72. Therefore, Wald confidence interval could not be computed for B3 and Clopper-Pearson Exact confidence interval is provided.
Time Frame: 72 weeks after the date of entry
Population: All participants with results expected at week 72
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Overall Study | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 448 | 234 | 61 | 62 | 6 | 54 | 31
proportion of participants | 0.64 [0.60 to 0.69] | 0.44 [0.37 to 0.50] | 0.92 [0.85 to 0.99] | 0.87 [0.79 to 0.95] | 1.00 [0.54 to 1.00] | 0.85 [0.76 to 0.95] | 0.77 [0.63 to 0.92]

4. Secondary Outcome: Number of Weeks of Follow-up
Description: All participants were followed on step 1/2 until 48 weeks after the last participant was enrolled to step 1 regardless of virologic status or treatment switches. Length of follow-up varied by Cohort.
Time Frame: From study entry through Step 1/2 follow-up
Population: all enrolled participants
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
weeks | 72 [60 to 96] | 96 [72 to 132] | 84 [72 to 126] | 96 [66 to 120] | 72 [60 to 96] | 96 [84 to 144]

5. Secondary Outcome: Time to Confirmed Virologic Failure, Defined as First HIV-1 RNA ≥1000 Copies/mL at or After 24 Weeks on Study
Description: Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure [specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry (to allow for 14 day window for scheduling the visit). HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement, allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure. Event times were the scheduled week of the initial failing measurement (RNA scheduled at week 0, 12, 24, 48 and every 24 weeks after). Censoring times were the scheduled week of the last RNA result. Length of follow-up varied by Cohort.
Time Frame: From week 24 through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
weeks
  1st percentile | 24 [24 to 24] | 24 [24 to 24] | 24 [24 to 72] | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | 24 [24 to 48] | 24 [24 to 24]
  5th percentile | 24 [24 to 24] | 48 [24 to NA] — Not estimable as the upper limit for survival function at all weeks is above 95% | 72 [24 to NA] — Not estimable as the upper limit for survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | 48 [24 to NA] — Not estimable as the upper limit for survival function at all weeks is above 95% | 24 [24 to 48]
  10th percentile | 24 [24 to 24] | NA [24 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 90% | 144 [48 to NA] — Not estimable as the upper limit for survival function at all weeks is above 90% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 90% | 120 [24 to NA] — Not estimable as the upper limit for survival function at all weeks is above 90% | 24 [24 to NA] — Not estimable as the upper limit for survival function at all weeks is above 90%
  25th percentile | 24 [24 to 24] | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 75% | NA [144 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 75% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 75% | NA [120 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 75% | NA [24 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 75%
  50th percentile | 60 [48 to 96] | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50% | NA [120 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 50% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50%

6. Secondary Outcome: Number of Participants With Confirmed Virologic Failure, Defined as First HIV-1 RNA ≥1000 Copies/mL at or After 24 Weeks on Study
Description: Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure [specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry (to allow for 14 day window for scheduling the visit). HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement, allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure. Length of follow-up varied by Cohort.
Time Frame: From week 24 through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
Participants | 145 | 6 | 4 | 0 | 5 | 6

7. Secondary Outcome: Percent of Participants With Confirmed Virologic Failure by Week 48
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure [specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry(to allow for 14 day window for scheduling the visit). HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement,allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure. Event times were the scheduled week of the initial failing measurement (RNA scheduled at week 0, 12, 24, 48 and every 24 weeks after). Censoring times were the scheduled week of the last RNA result. Length of follow-up varied by Cohort.
Time Frame: From week 24 to Week 48
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
percentage of participants | 48.9 [42.8 to 54.7] | 8.2 [3.3 to 16.0] | 2.9 [0.1 to 9.0] | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 5.8 [1.9 to 13.1] | 18.6 [7.4 to 33.8]

8. Secondary Outcome: Time to Confirmed Virologic Failure, Defined as First HIV-1 RNA ≥1000 Copies/mL at or After 24 Weeks on Study, With a New Resistance-associated Mutation Detected in Population-based Sequencing
Description: Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure [specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry (to allow for 14 day window for scheduling the visit). HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement, allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure. Event times were the scheduled week of the initial failing measurement (RNA scheduled at week 0, 12, 24, 48 and every 24 weeks after). Censoring times were the scheduled week of the last RNA result. Length of follow-up varied by Cohort. A new resistance-associated mutation is defined as one not present in the genotype prior to entry.
Time Frame: From week 24 through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
weeks
  1st percentile | 24 [24 to 24] | 24 [24 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99% | 24 [24 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | 48 [48 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99% | 24 [24 to 24]
  5th percentile | 24 [24 to 24] | NA [24 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 95% | NA [24 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [48 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 95% | 24 [24 to 48]
  10th percentile | 24 [24 to 48] | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 90% | NA [72 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 90% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 90% | NA [48 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 90% | 24 [24 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 90%
  25th percentile | 144 [72 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 75% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 75% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 75% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 75% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 75% | NA [24 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75%

9. Secondary Outcome: Number of Participants With Confirmed Virologic Failure, Defined as First HIV-1 RNA ≥1000 Copies/mL at or After 24 Weeks on Study, With a New Resistance-associated Mutation Detected in Population-based Sequencing
Description: Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure[specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry (to allow for 14 day window for scheduling the visit).HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement, allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure. Length of follow-up varied by Cohort. A new resistance-associated mutation is defined as one not present in the genotype prior to entry.
Time Frame: From week 24 through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
Participants | 48 | 1 | 2 | 0 | 1 | 5

10. Secondary Outcome: Percent of Participants With Confirmed Virologic Failure, Defined as First HIV-1 RNA ≥1000 Copies/mL at or After 24 Weeks on Study, With a New Resistance-associated Mutation Detected in Population-based Sequencing, by Week 48
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure[specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry(to allow for 14 day window for scheduling the visit).HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement,allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure.Event times were the scheduled week of the initial failing measurement(RNA scheduled at week 0, 12, 24, 48 and every 24 weeks after).Censoring times were the scheduled week of the last RNA result.Length of follow-up varied by Cohort.A new resistance-associated mutation is defined as one not present in the genotype prior to entry.
Time Frame: From week 24 to Week 48
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
percentage of participants | 16.6 [12.3 to 21.5] | 1.4 [0.1 to 6.6] | 1.4 [0.1 to 6.7] | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 1.5 [0.1 to 7.1] | 15.4 [5.5 to 29.9]

11. Secondary Outcome: Time From Study Entry/Randomization to Death
Description: Event time was the exact week of death. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit. Length of follow-up varied by Cohort.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
weeks
  1st percentile | 11.3 [4.0 to 17.7] | 3.1 [3.1 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99% | 44.6 [44.6 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | 77.9 [77.9 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99% | 2.4 [2.4 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99%
  5th percentile | 62.4 [17.7 to 110.1] | NA [3.1 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95% | NA [44.6 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [77.9 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95% | NA [2.4 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95%
  10th percentile | NA [82.1 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 90% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 90% | NA [51.4 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 90% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 90% | NA [77.9 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 90% | NA [2.4 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 90%

12. Secondary Outcome: Percent of Participants Experiencing Death by Week 48
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Event time was the exact week of death. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit.
Time Frame: From study entry to Week 48
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
percentage of participants | 3.9 [2.0 to 6.6] | 1.4 [0.1 to 6.5] | 1.4 [0.1 to 6.7] | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 2.9 [0.2 to 13.2]

13. Secondary Outcome: Time From Study Entry/Randomization to the First of Death, an AIDS-defining Event or a Non-AIDS-defining Event
Description: Event time was the exact week of death, AIDS-defining event or non-AIDS defining event. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit. Only new events were considered, an event that was also reported at or prior to study entry was not included. If a participant experienced multiple events, then the time of the first event was used in the analysis. AIDS defining events included parasitic, fungal, bacterial, and viral infections as well as neoplastic diseases, and neurological disorders. Non-AIDS defining events included malignancies, diabetes, neuropathies, cardiac and renal events. Length of follow-up varied by Cohort.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
weeks
  1st percentile | 4.0 [4.0 to 11.3] | 3.1 [3.1 to 34.0] | 16.3 [16.3 to 44.6] | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | 3.3 [3.3 to 26.6] | 2.4 [2.4 to 24.0]
  5th percentile | 27.6 [11.3 to 42.9] | 36.0 [3.1 to 84.0] | 50.3 [16.3 to 120.0] | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | 36.0 [3.3 to 119.1] | 24.0 [2.4 to 72.0]
  10th percentile | 57.9 [37.3 to 79.7] | 84.0 [4.6 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 90% | 120.0 [36.0 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 90% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 90% | 77.9 [3.6 to 142.4] | 48.4 [2.4 to 84.0]
  25th percentile | NA [118.6 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | NA [88.7 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | NA [120.0 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 75% | 142.4 [119.1 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 75% | 96.3 [48.4 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 75%

14. Secondary Outcome: Percent of Participants Experiencing Death, AIDS-defining Event or a Non-AIDS-defining Event by Week 48
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Event time was the exact week of death, AIDS-defining event or non-AIDS defining event. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit. Only new events were considered, an event that was also reported at or prior to study entry was not included. If a participant experienced multiple events, then the time of the first event was used in the analysis. AIDS defining events included parasitic, fungal, bacterial, and viral infections as well as neoplastic diseases, and neurological disorders. Non-AIDS defining events included malignancies, diabetes, neuropathies, cardiac and renal events.
Time Frame: From study entry to Week 48
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
percentage of participants | 8.8 [5.9 to 12.4] | 5.4 [1.7 to 12.2] | 4.2 [1.1 to 10.7] | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 5.8 [1.8 to 13.0] | 5.9 [1.0 to 17.4]

15. Secondary Outcome: Time From Study Entry/Randomization to the First of Death or Hospitalization.
Description: Event time was the exact week of death or hospitalization. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit. If a participant experienced multiple events, then the time of the first event was used in the analysis. Length of follow-up varied by Cohort.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
weeks
  1st percentile | 2.4 [1.0 to 5.9] | 2.3 [2.3 to 10.9] | 3.0 [3.0 to 25.6] | 16.4 [16.4 to 16.4] | 2.0 [2.0 to 3.3] | 2.3 [2.3 to 5.6]
  5th percentile | 13.4 [5.9 to 25.1] | 20.3 [2.3 to 100.1] | 28.0 [3.0 to 49.7] | 16.4 [16.4 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 95% | 7.7 [2.0 to 84.9] | 5.6 [2.3 to 96.1]
  10th percentile | 32.6 [22.9 to 61.1] | 80.7 [9.1 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 90% | 49.7 [6.1 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 90% | 16.4 [16.4 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 90% | 77.9 [2.0 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 90% | 96.1 [2.3 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 90%
  25th percentile | 120.1 [97.3 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 75% | NA [100.1 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | NA [90.7 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | NA [16.4 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | NA [84.9 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | NA [96.1 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75%
  50th percentile | 168.9 [168.9 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 50% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50% | NA [16.4 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 50% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50%

16. Secondary Outcome: Percent of Participants With Death or Hospitalization by Week 48
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Event time was the exact week of death or hospitalization. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit. If a participant experienced multiple events, then the time of the first event was used in the analysis.
Time Frame: From study entry to Week 48
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
percentage of participants | 12.3 [8.8 to 16.4] | 8.1 [3.3 to 15.8] | 9.7 [4.2 to 17.9] | 12.5 [0.5 to 44.5] | 5.7 [1.8 to 12.9] | 5.9 [1.0 to 17.4]

17. Secondary Outcome: Time From Study Entry/Randomization to Treatment Modification or Discontinuation.
Description: Treatment modification is defined as the first occurrence of a substitution or subtraction of one or more drugs in the study regimen, a temporary hold lasting 7 days or longer, or the addition of a new drug to the regimen. This would not include splitting any fixed dose combination medications if the participant continues on the active drugs of the combination. Event time was the exact week of the modification or discontinuation. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit. Length of follow-up varied by Cohort.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
weeks
  1st percentile | 1.0 [0.0 to 4.1] | 3.1 [3.1 to 28.9] | 4.4 [4.4 to 9.4] | 4.4 [4.4 to 4.4] | 0.1 [0.1 to 3.7] | 2.4 [2.4 to 5.1]
  5th percentile | 8.4 [4.1 to 18.9] | 33.4 [3.1 to 59.0] | 36.0 [4.4 to 38.6] | 4.4 [4.4 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 95% | 4.1 [0.1 to 29.7] | 5.1 [2.4 to 48.6]
  10th percentile | 25.3 [10.6 to 34.3] | 59.0 [15.0 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 90% | 38.6 [6.4 to 44.6] | 4.4 [4.4 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 90% | 29.7 [3.1 to 61.4] | 47.6 [2.4 to 55.0]
  25th percentile | 58.6 [48.1 to 84.0] | NA [117.6 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | 165.6 [43.0 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 75% | NA [4.4 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | NA [58.6 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | 98.9 [47.6 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 75%
  50th percentile | NA [120.7 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 50% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50% | NA [165.6 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 50% | NA [4.4 to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 50% | NA [98.9 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 50%

18. Secondary Outcome: Percent of Participants With Treatment Modification or Discontinuation by Week 48
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Treatment modification is defined as the first occurrence of a substitution or subtraction of one or more drugs in the study regimen, a temporary hold lasting 7 days or longer, or the addition of a new drug to the regimen. This would not include splitting any fixed dose combination medications if the participant continues on the active drugs of the combination. Event time was the exact week of the modification or discontinuation. Censoring time was the earliest time point between last dose week and the week of the last step 1/2 visit.
Time Frame: From study entry to Week 48
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
percentage of participants | 19.9 [15.5 to 24.7] | 6.8 [2.5 to 14.0] | 19.4 [11.2 to 29.3] | 12.5 [0.5 to 44.5] | 14.3 [7.3 to 23.6] | 11.8 [3.6 to 25.1]

19. Secondary Outcome: Time From Study Entry/Randomization to Treatment Modification or Discontinuation Due to Toxicity
Description: Treatment modification is defined as the first occurrence of a substitution or subtraction of one or more drugs in the study regimen, a temporary hold lasting 7 days or longer, or the addition of a new drug to the regimen, due to an adverse event. This would not include splitting any fixed dose combination medications if the participant continues on the active drugs of the combination. Event time was the exact week of the modification or discontinuation. Censoring time was the earliest time point between last dose week and the week of the last step 1/2 visit. Length of follow-up varied by Cohort. DAIDS AE Grading Table, Version 1.0 was used.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
weeks
  1st percentile | 2.1 [0.4 to 32.3] | 15.0 [15.0 to 49.1] | 6.4 [6.4 to 134.0] | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | 0.1 [0.1 to 3.7] | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99%
  5th percentile | 106.1 [32.3 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 95% | NA [15.0 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95% | 134.0 [6.4 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [0.1 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95%
  10th percentile | NA [106.1 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 90% | NA [41 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 90% | NA [134.0 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 90% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 90% | NA [3.1 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 90% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 90%

20. Secondary Outcome: Percent of Participants With Treatment Modification or Discontinuation Due to Toxicity by Week 48
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Treatment modification is defined as the first occurrence of a substitution or subtraction of one or more drugs in the study regimen, a temporary hold lasting 7 days or longer, or the addition of a new drug to the regimen, due to an adverse event. This would not include splitting any fixed dose combination medications if the participant continues on the active drugs of the combination. Event time was the exact week of the modification or discontinuation. Censoring time was the earliest time point between last dose week and the week of the last step 1/2 visit. DAIDS AE Grading Table, Version 1.0 was used.
Time Frame: From study entry to Week 48
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
percentage of participants | 3.2 [1.6 to 5.8] | 2.7 [0.5 to 8.6] | 1.4 [0.1 to 6.7] | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 4.3 [1.1 to 11.0] | 0 [NA to NA] — Not estimated due to lack of events in group by week 48

21. Secondary Outcome: Time From Study Entry/Randomization to the Development of Immune Reconstitution Inflammatory Syndrome (IRIS)
Description: Event time was the exact week of the diagnosis. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit. Length of follow-up varied by Cohort.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
weeks
  1st percentile | NA [9.0 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 99% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | 25.0 [25.0 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | 13.0 [13.0 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99%
  5th percentile | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [25.0 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [13.0 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95%

22. Secondary Outcome: Percent of Participants That Developed Immune Reconstitution Inflammatory Syndrome (IRIS) by Week 48
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Event time was the exact week of the diagnosis. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit.
Time Frame: From study entry to week 48
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
percentage of participants | 0.7 [0.1 to 2.4] | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 1.4 [0.1 to 6.7] | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 3.0 [0.2 to 13.6]

23. Secondary Outcome: Time to First Dose Modification Due to Grade 3 or 4 Toxicity
Description: Event time was the exact week of the modification. Censoring time was the earliest time point between last dose week and the week of the last step 1/2 visit. Length of follow-up varied by Cohort. DAIDS AE Grading Table, Version 1.0 was used.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
weeks
  1st percentile | 45.7 [5.9 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99% | 63.3 [63.3 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 99%
  5th percentile | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [63.3 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95%

24. Secondary Outcome: Percent of Participants With a Dose Modification Due to Grade 3 or 4 Toxicity by Week 48
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Event time was the exact week of the modification. Censoring time was the earliest time point between last dose week and the week of the last step 1/2 visit. DAIDS AE Grading Table, Version 1.0 was used.
Time Frame: From study entry to week 48
Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
percentage of participants | 1.0 [0.3 to 2.8] | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 0 [NA to NA] — Not estimated due to lack of events in group by week 48 | 0 [NA to NA] — Not estimated due to lack of events in group by week 48

25. Secondary Outcome: Change From Baseline in CD4+ T-cell Count
Description: Baseline is defined as the last measurement obtained on or before the earlier of the following two dates: the date of entry/randomization plus three days (this is the time allowed in the protocol for starting study-defined ART) and the date of starting the study-defined ARV regimen (this second date applies only to Cohorts B, C and D as there is no change of regimen for patients in Cohort A)
Time Frame: Baseline, week 24, 48, and 72
Population: all enrolled participants with results available at baseline and at the given follow-up time point
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
cells/mm^3
  Change from baseline at week 24: number analyzed (Participants) | 267 | 70 | 71 | 8 | 69 | 33
  Change from baseline at week 24 | 39 (105) | 109 (133) | 116 (130) | 142 (99) | 100 (121) | 90 (131)
  Change from baseline at week 48: number analyzed (Participants) | 258 | 71 | 68 | 8 | 69 | 31
  Change from baseline at week 48 | 65 (138) | 157 (162) | 158 (172) | 86 (166) | 160 (140) | 135 (214)
  Change from baseline at week 72: number analyzed (Participants) | 207 | 59 | 58 | 6 | 52 | 30
  Change from baseline at week 72 | 87 (165) | 182 (153) | 197 (199) | 238 (86) | 185 (151) | 165 (270)

26. Secondary Outcome: Change From Baseline in Fasting Values of Total Cholesterol
Description: as for outcome 25
Time Frame: Baseline, week 24, 48 and 72
Population: all enrolled participants with results available at baseline and at the given follow-up time point
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
mg/dL
  Change from baseline at week 24: number analyzed (Participants) | 195 | 50 | 51 | 6 | 54 | 25
  Change from baseline at week 24 | 5.7 (33.0) | 16.7 (41.8) | 32.5 (43.3) | 12.4 (27.5) | 16.5 (36.5) | 7.9 (43.5)
  Change from baseline at week 48: number analyzed (Participants) | 189 | 54 | 48 | 6 | 57 | 22
  Change from baseline at week 48 | 4.4 (36.0) | 19.7 (41.1) | 40.4 (46.9) | 9.9 (21.6) | 20.0 (34.6) | 19.1 (32.0)
  Change from baseline at week 72: number analyzed (Participants) | 149 | 41 | 42 | 5 | 43 | 20
  Change from baseline at week 72 | 7.6 (33.4) | 22.6 (47.8) | 40.4 (51.0) | 28.2 (42.9) | 22.1 (35.5) | 24.5 (33.9)

27. Secondary Outcome: Change From Baseline in Fasting Values of High-density Lipoprotein Cholesterol
Description: Baseline is defined as the last measurement obtained on or before the earlier of the following two dates: the date of entry/randomization plus three days (this is the time allowed in the protocol for starting study-defined ART) and the date of starting the study-defined ARV regimen (this second date applies only to Cohorts B, C and D as there is no change of regimen for patients in Cohort A)]
Time Frame: Baseline, week 24, 48 and 72
Population: all enrolled participants with results available at baseline and at the given follow-up time point
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
mg/dL
  Change from baseline at week 24: number analyzed (Participants) | 181 | 48 | 49 | 6 | 54 | 24
  Change from baseline at week 24 | 2.8 (14.7) | 3.2 (11.7) | 11.4 (16.8) | 2.1 (4.3) | 1.0 (13.2) | -2.2 (11.3)
  Change from baseline at week 48: number analyzed (Participants) | 183 | 53 | 47 | 6 | 58 | 23
  Change from baseline at week 48 | 3.5 (13.9) | 5.3 (10.3) | 13.4 (13.8) | 3.8 (2.9) | 2.3 (12.2) | 1.8 (12.2)
  Change from baseline at week 72: number analyzed (Participants) | 143 | 39 | 41 | 5 | 43 | 19
  Change from baseline at week 72 | 4.7 (14.1) | 4.4 (11.4) | 15.7 (15.1) | 4.6 (3.6) | 5.8 (13.2) | 3.4 (12.8)

28. Secondary Outcome: Change From Baseline in Fasting Values of Calculated Low-density Lipoprotein Cholesterol
Description: as for outcome 25
Time Frame: Baseline, week 24, 48 and 72
Population: all enrolled participants with results available at baseline and at the given follow-up time point
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
mg/dL
  Change from baseline at week 24: number analyzed (Participants) | 193 | 48 | 51 | 6 | 52 | 24
  Change from baseline at week 24 | 1.3 (25.2) | 13.3 (34.4) | 21.5 (31.6) | -0.5 (11.3) | 12.2 (25.4) | 9.9 (26.9)
  Change from baseline at week 48: number analyzed (Participants) | 185 | 51 | 45 | 7 | 56 | 22
  Change from baseline at week 48 | 3.4 (28.5) | 16.3 (32.8) | 28.2 (38.1) | 0.3 (17.0) | 15.3 (25.7) | 14.4 (25.2)
  Change from baseline at week 72: number analyzed (Participants) | 148 | 39 | 39 | 5 | 42 | 18
  Change from baseline at week 72 | 3.9 (26.6) | 22.4 (38.6) | 27.8 (40.1) | 16.6 (37.2) | 13.6 (25.8) | 19.7 (27.4)

29. Secondary Outcome: Change From Baseline in Fasting Values of Triglycerides
Description: as for outcome 25
Time Frame: Baseline, week 24, 48 and 72
Population: all enrolled participants with results available at baseline and at the given follow-up time point
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
mg/dL
  Change from baseline at week 24: number analyzed (Participants) | 192 | 47 | 53 | 6 | 50 | 24
  Change from baseline at week 24 | 15.4 (75.7) | -3.6 (84.9) | 27.6 (112.5) | 36.0 (48.1) | 15.4 (84.4) | 28.9 (65.5)
  Change from baseline at week 48: number analyzed (Participants) | 184 | 53 | 49 | 6 | 53 | 23
  Change from baseline at week 48 | 12.2 (70.8) | -11.5 (136.7) | 19.9 (84.1) | 22.2 (57.2) | 9.9 (65.9) | 24.4 (90.1)
  Change from baseline at week 72: number analyzed (Participants) | 144 | 40 | 43 | 5 | 41 | 22
  Change from baseline at week 72 | 17.5 (79.1) | -31.3 (122.3) | 18.9 (99.4) | 20.7 (56.3) | 11.8 (83.9) | 6.7 (71.1)

30. Secondary Outcome: Change From Baseline in Fasting Values of Glucose
Description: as for outcome 25
Time Frame: Baseline, week 24, 48 and 72
Population: all enrolled participants with results available at baseline and at the given follow-up time point
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
Number analyzed (Participants) | 287 | 74 | 72 | 8 | 70 | 34
mg/dL
  Change from baseline at week 24: number analyzed (Participants) | 195 | 49 | 51 | 5 | 52 | 27
  Change from baseline at week 24 | 1.9 (25.0) | 8.8 (18.9) | 6.1 (22.3) | 6.6 (8.3) | 2.1 (19.9) | 3.2 (19.1)
  Change from baseline at week 48: number analyzed (Participants) | 183 | 55 | 49 | 5 | 55 | 25
  Change from baseline at week 48 | 2.1 (19.8) | 9.3 (28.5) | 6.2 (20.1) | 1.7 (6.9) | 3.0 (16.7) | 4.2 (13.7)
  Change from baseline at week 72: number analyzed (Participants) | 146 | 42 | 43 | 4 | 43 | 23
  Change from baseline at week 72 | 3.0 (29.7) | 6.8 (23.8) | -5.2 (79.1) | 4.3 (7.6) | -0.9 (17.9) | 7.8 (13.7)

31. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA ≤200 Copies/mL at 48 Weeks [CPI+SOC v SOC]
Description: The measurement closest to exactly 48 weeks (ie, 7x48=336 days) after the date of entry, within the window of 48 weeks ± 6 weeks (specifically 295 to 378 days after randomization, inclusive).
  The analysis in the protocol and in the Stat. Analysis Plan involved estimating the proportion of participants in the overall study population with HIV-1 RNA ≤200 copies/mL at week 48 with a 95% confidence interval calculated via a Wald approach. Death or lost to follow-up before week 48 was considered as HIV-1 RNA>200 copies/mL at week 48. Missing results at week 48 were considered as HIV-1 RNA >200 copies/mL at week 48 unless the immediately preceding and succeeding HIV-1 RNA measurements were ≤200 copies/mL.
Time Frame: 48 weeks after the date of entry
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
proportion of participants | 0.66 [0.60 to 0.72] | 0.62 [0.56 to 0.68]

32. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA ≤200 Copies/mL at 24 Weeks [CPI+SOC v SOC]
Description: The measurement closest to exactly 24 weeks (ie, 7x24=168 days) after the date of entry, within the window of 24 weeks ± 6 weeks (specifically 127 to 210 days after randomization, inclusive).
  The analysis in the protocol and in the Stat. Analysis Plan involved estimating the proportion of participants in the overall study population with HIV-1 RNA ≤200 copies/mL at week 24 with a 95% confidence interval calculated via a Wald approach. Death or lost to follow-up before week 24 was considered as HIV-1 RNA>200 copies/mL at week 24. Missing results at week 24 were considered as HIV-1 RNA >200 copies/mL at week 24 unless the immediately preceding and succeeding HIV-1 RNA measurements were ≤200 copies/mL.
Time Frame: 24 weeks after the date of entry
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
proportion of participants | 0.68 [0.62 to 0.73] | 0.61 [0.55 to 0.67]

33. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA ≤200 Copies/mL at 72 Weeks [CPI+SOC v SOC]
Description: The measurement closest to exactly 72 weeks (ie, 7x72=504 days) after the date of entry, within the window of 72 weeks ± 6 weeks (specifically 463 to 546 days, inclusive).
  The analysis in the protocol and in the Analysis Plan involved estimating the proportion of participants in the overall study population with HIV-1 RNA ≤200 copies/mL at week 72 with a 95% confidence interval calculated via a Wald approach. Death or lost to follow-up before week 72 was considered as HIV-1 RNA>200 copies/mL at week 72. If a result was expected, missing results at week 72 were considered as HIV-1 RNA >200 copies/mL at week 72 unless the immediately preceding and succeeding HIV-1 RNA measurements were ≤200 copies/mL.
Time Frame: 72 weeks after the date of entry
Population: All participants randomized to either CPI+SOC or SOC with results expected at week 72
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 210 | 217
proportion of participants | 0.69 [0.62 to 0.75] | 0.62 [0.55 to 0.68]

34. Secondary Outcome: Number of Weeks of Follow-up [CPI+SOC v SOC]
Description: All participants were followed on step 1/2 until 48 weeks after the last participant was enrolled to step 1 regardless of virologic status or treatment switches.
Time Frame: From study entry through Step 1/2 follow-up
Population: All participants randomized to either CPI+SOC or SOC
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
weeks | 72 [72 to 108] | 72 [72 to 108]

35. Secondary Outcome: Time to Confirmed Virologic Failure, Defined as First HIV-1 RNA ≥1000 Copies/mL at or After 24 Weeks on Study [CPI+SOC v SOC]
Description: Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure [specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry (to allow for 14 day window for scheduling the visit). HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement, allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure. Event times were the scheduled week of the initial failing measurement (RNA scheduled at week 0, 12, 24, 48 and every 24 weeks after). Censoring times were the scheduled week of the last RNA result.
Time Frame: From week 24 through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
weeks
  1st percentile | 24 [24 to 24] | 24 [24 to 24]
  5th percentile | 24 [24 to 24] | 24 [24 to 24]
  10th percentile | 24 [24 to 24] | 24 [24 to 24]
  25th percentile | 60 [48 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75% | 24 [24 to 48]
  50th percentile | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for survival function at all weeks is above 50% | NA [144 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 50%

36. Secondary Outcome: Number of Participants With Confirmed Virologic Failure, Defined as First HIV-1 RNA ≥1000 Copies/mL at or After 24 Weeks on Study [CPI+SOC v SOC]
Description: Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure [specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry (to allow for 14 day window for scheduling the visit). HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement, allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure.
Time Frame: From week 24 through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Count of Participants; unit: Participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
Participants | 66 | 89

37. Secondary Outcome: Percent of Participants With Confirmed Virologic Failure by Week 48 [CPI+SOC v SOC]
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure [specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry(to allow for 14 day window for scheduling the visit). HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement,allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure. Event times were the scheduled week of the initial failing measurement (RNA scheduled at week 0, 12, 24, 48 and every 24 weeks after). Censoring times were the scheduled week of the last RNA result.
Time Frame: From week 24 to Week 48
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
percentage of participants | 24.9 [19.6 to 30.4] | 32.2 [26.6 to 37.9]

38. Secondary Outcome: Time to Confirmed Virologic Failure, Defined as First HIV-1 RNA ≥1000 Copies/mL at or After 24 Weeks on Study, With a New Resistance-associated Mutation Detected in Population-based Sequencing [CPI+SOC v SOC]
Description: Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure [specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry (to allow for 14 day window for scheduling the visit). HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement, allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure. Event times were the scheduled week of the initial failing measurement (RNA scheduled at week 0, 12, 24, 48 and every 24 weeks after). Censoring times were the scheduled week of the last RNA result. A new resistance-associated mutation is defined as one not present in the genotype prior to entry.
Time Frame: From week 24 through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
weeks
  1st percentile | 24 [24 to 24] | 24 [24 to 24]
  5th percentile | 24 [24 to 48] | 24 [24 to 24]
  10th percentile | NA [24 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 90% | 48 [24 to 144]
  25th percentile | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 75% | NA [144 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75%

39. Secondary Outcome: Number of Participants With Confirmed Virologic Failure, Defined as First HIV-1 RNA ≥1000 Copies/mL at or After 24 Weeks on Study, With a New Resistance-associated Mutation Detected in Population-based Sequencing [CPI+SOC v SOC]
Description: Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure[specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry (to allow for 14 day window for scheduling the visit).HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement, allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure. A new resistance-associated mutation is defined as one not present in the genotype prior to entry.
Time Frame: From week 24 through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Count of Participants; unit: Participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
Participants | 20 | 32

40. Secondary Outcome: Percent of Participants With Confirmed Virologic Failure, Defined as First HIV-1 RNA ≥1000 Copies/mL at or After 24 Weeks on Study, With a New Resistance-associated Mutation Detected in Population-based Sequencing, by Week 48 [CPI+SOC v SOC]
Description: Results report percent of participants reaching outcome by week 48 using Kaplan-Meier method. Virologic failure was confirmed by the next HIV-1 RNA measurement ≥1000 copies/mL (irrespective of time between initial and confirmatory measure[specimens on separate dates] and treatment status). A week 24 measurement included HIV-1 RNA obtained ≥7*22=154 days after study entry(to allow for 14 day window for scheduling the visit).HIV-1 RNA measurements through and including 21 November 2016 were considered in identifying an initial failing measurement,allowing HIV-1 RNA at the close-out visit between 22 November 2016 and 13 February 2017 to be a confirmatory measure.Event times were the scheduled week of the initial failing measurement(RNA scheduled at week 0, 12, 24, 48 and every 24 weeks after).Censoring times were the scheduled week of the last RNA result.A new resistance-associated mutation is defined as one not present in the genotype prior to entry.
Time Frame: From week 24 to Week 48
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
percentage of participants | 7.8 [4.9 to 11.7] | 12.1 [8.4 to 16.6]

41. Secondary Outcome: Time From Study Entry/Randomization to Death [CPI+SOC v SOC]
Description: Event time was the exact week of death. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
weeks
  1st percentile | 11.3 [3.1 to 27.4] | 15.9 [2.4 to 51.4]
  5th percentile | NA [27.4 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95% | 82.1 [51.4 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 95%
  10th percentile | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 90% | NA [110.1 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 90%

42. Secondary Outcome: Percent of Participants Experiencing Death by Week 48 [CPI+SOC v SOC]
Description: as for outcome 12
Time Frame: From study entry to Week 48
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
percentage of participants | 3.9 [2.0 to 6.8] | 1.5 [0.5 to 3.6]

43. Secondary Outcome: Time From Study Entry/Randomization to the First of Death, an AIDS-defining Event or a Non-AIDS-defining Event [CPI+SOC v SOC]
Description: Event time was the exact week of death, AIDS-defining event or non-AIDS defining event. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit. Only new events were considered, an event that was also reported at or prior to study entry was not included. If a participant experienced multiple events, then the time of the first event was used in the analysis. AIDS defining events included parasitic, fungal, bacterial, and viral infections as well as neoplastic diseases, and neurological disorders. Non-AIDS defining events included malignancies, diabetes, neuropathies, cardiac and renal events.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
weeks
  1st percentile | 4.0 [3.1 to 4.0] | 4.0 [2.4 to 12.0]
  5th percentile | 27.6 [4.0 to 42.9] | 42.3 [12.4 to 58.9]
  10th percentile | 60.6 [36.0 to 84.0] | 77.9 [48.0 to 91.6]
  25th percentile | NA [142.4 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75% | NA [112.7 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75%

44. Secondary Outcome: Percent of Participants Experiencing Death, AIDS-defining Event or a Non-AIDS-defining Event by Week 48 [CPI+SOC v SOC]
Description: as for outcome 14
Time Frame: From study entry to Week 48
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
percentage of participants | 8.2 [5.3 to 12.0] | 6.5 [3.9 to 9.9]

45. Secondary Outcome: Time From Study Entry/Randomization to the First of Death or Hospitalization [CPI+SOC v SOC]
Description: Event time was the exact week of death or hospitalization. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit. If a participant experienced multiple events, then the time of the first event was used in the analysis.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
weeks
  1st percentile | 2.3 [2.0 to 4.0] | 2.3 [1.0 to 5.6]
  5th percentile | 11.3 [4.0 to 25.1] | 20.3 [8.7 to 32.4]
  10th percentile | 44.6 [20.6 to 90.7] | 45.3 [25.6 to 77.9]
  25th percentile | 168.9 [119.6 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 75% | NA [107.3 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 75%

46. Secondary Outcome: Percent of Participants With Death or Hospitalization by Week 48 [CPI+SOC v SOC]
Description: as for outcome 16
Time Frame: From study entry to Week 48
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
percentage of participants | 10.6 [7.2 to 14.7] | 10.6 [7.3 to 14.7]

47. Secondary Outcome: Time From Study Entry/Randomization to Treatment Modification or Discontinuation [CPI+SOC v SOC]
Description: Treatment modification is defined as the first occurrence of a substitution or subtraction of one or more drugs in the study regimen, a temporary hold lasting 7 days or longer, or the addition of a new drug to the regimen. This would not include splitting any fixed dose combination medications if the participant continues on the active drugs of the combination. Event time was the exact week of the modification or discontinuation. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
weeks
  1st percentile | 1.0 [0.0 to 3.7] | 2.4 [0.1 to 5.9]
  5th percentile | 5.1 [3.7 to 9.3] | 22.3 [9.0 to 31.9]
  10th percentile | 23.6 [6.9 to 36.0] | 38.9 [26.0 to 47.0]
  25th percentile | 84.0 [48.7 to 148.3] | 111.1 [72.4 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 75%

48. Secondary Outcome: Percent of Participants With Treatment Modification or Discontinuation by Week 48 [CPI+SOC v SOC]
Description: as for outcome 18
Time Frame: From study entry to Week 48
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
percentage of participants | 19.1 [14.5 to 24.1] | 13.6 [9.8 to 18.1]

49. Secondary Outcome: Time From Study Entry/Randomization to Treatment Modification or Discontinuation Due to Toxicity [CPI+SOC v SOC]
Description: Treatment modification is defined as the first occurrence of a substitution or subtraction of one or more drugs in the study regimen, a temporary hold lasting 7 days or longer, or the addition of a new drug to the regimen, due to an adverse event. This would not include splitting any fixed dose combination medications if the participant continues on the active drugs of the combination. Event time was the exact week of the modification or discontinuation. Censoring time was the earliest time point between last dose week and the week of the last step 1/2 visit. DAIDS AE Grading Table, Version 1.0 was used.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
weeks
  1st percentile | 3.1 [0.4 to 5.0] | 9.0 [0.1 to 41.0]
  5th percentile | NA [5.0 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95% | NA [41.0 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95%

50. Secondary Outcome: Percent of Participants With Treatment Modification or Discontinuation Due to Toxicity by Week 48 [CPI+SOC v SOC]
Description: as for outcome 20
Time Frame: From study entry to Week 48
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
percentage of participants | 2.8 [1.2 to 5.3] | 2.3 [1.0 to 4.7]

51. Secondary Outcome: Time From Study Entry/Randomization to the Development of Immune Reconstitution Inflammatory Syndrome (IRIS) [CPI+SOC v SOC]
Description: Event time was the exact week of the diagnosis. Censoring time was the earlier of last contact week and the week of the last step 1/2 visit.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
weeks
  1st percentile | NA [9.0 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 99% | 25.0 [13.0 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 99%
  5th percentile | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95%

52. Secondary Outcome: Percent of Participants That Developed Immune Reconstitution Inflammatory Syndrome (IRIS) by Week 48 [CPI+SOC v SOC]
Description: as for outcome 22
Time Frame: From study entry to Week 48
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
percentage of participants | 0.4 [.03 to 2.1] | 1.1 [0.3 to 3.1]

53. Secondary Outcome: Time to First Dose Modification Due to Grade 3 or 4 Toxicity [CPI+SOC v SOC]
Description: Event time was the exact week of the modification. Censoring time was the earliest time point between last dose week and the week of the last step 1/2 visit. DAIDS AE Grading Table, Version 1.0 was used.
Time Frame: From study entry through Step 1/2 follow-up; median (IQR) step 1/2 follow-up was 72 (72,108) weeks
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
weeks
  1st percentile | 45.7 [5.9 to NA] — Not estimable as the upper limit for the survival function at all weeks is above 95% | NA [63.3 to NA] — Not estimable as the estimate and upper limit for the survival function at all weeks is above 95%
  5th percentile | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95% | NA [NA to NA] — Not estimable as the estimate, lower limit and upper limit for the survival function at all weeks is above 95%

54. Secondary Outcome: Percent of Participants With a Dose Modification Due to Grade 3 or 4 Toxicity by Week 48 [CPI+SOC v SOC]
Description: as for outcome 24
Time Frame: From study entry to Week 48
Population: All participants randomized to either CPI+SOC or SOC
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
percentage of participants | 1.2 [0.3 to 3.2] | 0 [NA to NA] — Not estimated due to lack of events in group by week 48

55. Secondary Outcome: Change From Baseline in CD4+ T-cell Count [CPI+SOC v SOC]
Description: Baseline is defined as the last measurement obtained on or before the earlier of the following two dates: the date of entry/randomization plus three days (this is the time allowed in the protocol for starting study-defined ART) and the date of starting the study-defined ARV regimen.
Time Frame: Baseline, week 24, 48, and 72
Population: All participants randomized to either CPI+SOC or SOC with results available at baseline and at the given follow-up time point
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
cells/mm^3
  Change from baseline at week 24: number analyzed (Participants) | 241 | 254
  Change from baseline at week 24 | 72 (125) | 74 (118)
  Change from baseline at week 48: number analyzed (Participants) | 235 | 247
  Change from baseline at week 48 | 112 (162) | 107 (157)
  Change from baseline at week 72: number analyzed (Participants) | 193 | 199
  Change from baseline at week 72 | 145 (195) | 134 (170)

56. Secondary Outcome: Change From Baseline in Fasting Values of Total Cholesterol [CPI+SOC v SOC]
Description: as for outcome 55
Time Frame: Baseline, week 24, 48, and 72
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
mg/dL
  Change from baseline at week 24: number analyzed (Participants) | 183 | 183
  Change from baseline at week 24 | 10.1 (37.4) | 14.4 (38.8)
  Change from baseline at week 48: number analyzed (Participants) | 181 | 181
  Change from baseline at week 48 | 15.1 (39.1) | 14.1 (40.6)
  Change from baseline at week 72: number analyzed (Participants) | 145 | 144
  Change from baseline at week 72 | 17.4 (41.8) | 18.7 (40.2)

57. Secondary Outcome: Change From Baseline in Fasting Values of High-density Lipoprotein Cholesterol [CPI+SOC v SOC]
Description: as for outcome 55
Time Frame: Baseline, week 24, 48, and 72
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
mg/dL
  Change from baseline at week 24: number analyzed (Participants) | 174 | 175
  Change from baseline at week 24 | 2.9 (13.0) | 3.6 (16.1)
  Change from baseline at week 48: number analyzed (Participants) | 176 | 179
  Change from baseline at week 48 | 5.6 (12.6) | 3.7 (14.3)
  Change from baseline at week 72: number analyzed (Participants) | 141 | 139
  Change from baseline at week 72 | 6.0 (13.7) | 6.6 (14.7)

58. Secondary Outcome: Change From Baseline in Fasting Values of Calculated Low-density Lipoprotein Cholesterol [CPI+SOC v SOC]
Description: as for outcome 55
Time Frame: Baseline, week 24, 48, and 72
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
mg/dL
  Change from baseline at week 24: number analyzed (Participants) | 178 | 181
  Change from baseline at week 24 | 5.5 (29.9) | 9.5 (27.0)
  Change from baseline at week 48: number analyzed (Participants) | 176 | 176
  Change from baseline at week 48 | 12.0 (31.9) | 10.1 (30.0)
  Change from baseline at week 72: number analyzed (Participants) | 142 | 138
  Change from baseline at week 72 | 11.9 (33.3) | 12.8 (31.2)

59. Secondary Outcome: Change From Baseline in Fasting Values of Triglycerides [CPI+SOC v SOC]
Description: as for outcome 55
Time Frame: Baseline, week 24, 48, and 72
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
mg/dL
  Change from baseline at week 24: number analyzed (Participants) | 177 | 180
  Change from baseline at week 24 | 15.3 (86.9) | 18.7 (80.4)
  Change from baseline at week 48: number analyzed (Participants) | 178 | 175
  Change from baseline at week 48 | 2.2 (89.4) | 19.6 (81.1)
  Change from baseline at week 72: number analyzed (Participants) | 144 | 140
  Change from baseline at week 72 | 13.7 (103.4) | 7.1 (73.7)

60. Secondary Outcome: Change From Baseline in Fasting Values of Glucose [CPI+SOC v SOC]
Description: as for outcome 55
Time Frame: Baseline, week 24, 48, and 72
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cell Phone Intervention (CPI) + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 257 | 264
mg/dL
  Change from baseline at week 24: number analyzed (Participants) | 178 | 184
  Change from baseline at week 24 | 3.7 (26.1) | 3.7 (18.2)
  Change from baseline at week 48: number analyzed (Participants) | 172 | 185
  Change from baseline at week 48 | 3.6 (16.5) | 5.1 (23.1)
  Change from baseline at week 72: number analyzed (Participants) | 141 | 148
  Change from baseline at week 72 | 3.6 (29.0) | 1.5 (45.9)

ADVERSE EVENTS:
Time Frame: From enrollment to the end of step 1/2 follow up. Participants were followed in Steps 1 and 2 until 48 weeks after the last participant was enrolled to Step 1. Median follow-up time was 72 weeks, maximum of 204 weeks.
Description: Version 2.0 of the DAIDS EAE Manual was used for this study. At entry, signs, symptoms and laboratory values regardless of grade that occurred <30 days before entry were reported. Post-entry, signs/symptoms and laboratory values grade ≥3, or caused a change in treatment/ART regardless of grade, were reported. Diagnoses identified on the study-specific list, or caused a change in treatment, were recorded at all visits. Used DAIDS AE Grading Table, Version 1.0, December 2004 (clarified AUG09)
Arm/Group | Experimental: Cohort A | Experimental: Sub-cohort B1 | Experimental: Sub-cohort B2 | Experimental: Sub-cohort B3 | Experimental: Cohort C | Experimental: Cohort D
All-Cause Mortality (participants affected / at risk) | 18/287 | 1/74 | 2/72 | 0/8 | 1/70 | 1/34
Serious Adverse Events (participants affected / at risk) | 61/287 | 8/74 | 13/72 | 1/8 | 9/70 | 6/34
Other Adverse Events (participants affected / at risk) | 283/287 | 72/74 | 69/72 | 8/8 | 69/70 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Cohort A (N=287) | Experimental: Sub-cohort B1 (N=74) | Experimental: Sub-cohort B2 (N=72) | Experimental: Sub-cohort B3 (N=8) | Experimental: Cohort C (N=70) | Experimental: Cohort D (N=34)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0 | 1
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 3 | 0 | 0 | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Immunosuppression (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Amoebiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 4 | 0 | 1 | 0 | 1 | 0
Cerebral toxoplasmosis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 2 | 0 | 0 | 0 | 0
HIV-associated neurocognitive disorder (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Leptospirosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 1
Meningitis pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Neurocryptococcosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Scrub typhus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dystonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 5 | 1 | 1 | 0 | 2 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Cohort A (N=287) | Experimental: Sub-cohort B1 (N=74) | Experimental: Sub-cohort B2 (N=72) | Experimental: Sub-cohort B3 (N=8) | Experimental: Cohort C (N=70) | Experimental: Cohort D (N=34)
Conjunctivitis allergic (Eye disorders) | 1 | 2 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 2 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 18 | 3 | 5 | 0 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 7 | 1 | 3 | 0 | 1 | 2
Abdominal tenderness (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 22 | 6 | 7 | 0 | 0 | 3
Peptic ulcer (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 23 | 2 | 3 | 0 | 3 | 1
Chest pain (General disorders) | 10 | 1 | 2 | 1 | 0 | 0
Chills (General disorders) | 3 | 1 | 4 | 1 | 0 | 2
Fatigue (General disorders) | 5 | 2 | 4 | 1 | 1 | 0
Oedema peripheral (General disorders) | 2 | 0 | 1 | 0 | 0 | 2
Pain (General disorders) | 2 | 3 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 53 | 8 | 8 | 2 | 8 | 9
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 2 | 1 | 1 | 0 | 1 | 2
Acute sinusitis (Infections and infestations) | 6 | 1 | 2 | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 3
Bacterial vaginosis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 3
Body tinea (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 3
Chronic hepatitis B (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 5 | 1 | 4 | 0 | 0 | 2
Helminthic infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 9 | 3 | 3 | 0 | 4 | 0
Influenza (Infections and infestations) | 3 | 1 | 2 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 19 | 1 | 2 | 0 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 11 | 1 | 0 | 0 | 2 | 2
Purulent discharge (Infections and infestations) | 4 | 2 | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 19 | 2 | 7 | 2 | 6 | 3
Urinary tract infection (Infections and infestations) | 15 | 7 | 0 | 1 | 2 | 3
Vulvovaginal candidiasis (Infections and infestations) | 7 | 4 | 2 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 41 | 12 | 6 | 1 | 11 | 6
Aspartate aminotransferase increased (Investigations) | 68 | 14 | 13 | 2 | 18 | 8
Blood alkaline phosphatase abnormal (Investigations) | 1 | 1 | 0 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 68 | 20 | 16 | 1 | 26 | 7
Blood bicarbonate decreased (Investigations) | 94 | 22 | 23 | 3 | 27 | 14
Blood bilirubin increased (Investigations) | 106 | 19 | 12 | 3 | 22 | 6
Blood cholesterol increased (Investigations) | 65 | 41 | 40 | 3 | 31 | 16
Blood creatinine increased (Investigations) | 37 | 10 | 8 | 1 | 9 | 4
Blood glucose decreased (Investigations) | 32 | 6 | 10 | 0 | 7 | 0
Blood glucose increased (Investigations) | 72 | 15 | 22 | 0 | 21 | 11
Blood phosphorus decreased (Investigations) | 75 | 25 | 21 | 1 | 20 | 12
Blood potassium decreased (Investigations) | 34 | 12 | 4 | 0 | 4 | 5
Blood potassium increased (Investigations) | 14 | 0 | 4 | 1 | 5 | 0
Blood pressure increased (Investigations) | 6 | 2 | 1 | 0 | 1 | 2
Blood sodium decreased (Investigations) | 145 | 44 | 32 | 8 | 42 | 16
Blood sodium increased (Investigations) | 42 | 4 | 7 | 1 | 4 | 2
Blood triglycerides increased (Investigations) | 8 | 6 | 5 | 0 | 3 | 2
Haemoglobin decreased (Investigations) | 40 | 8 | 9 | 2 | 6 | 7
Low density lipoprotein increased (Investigations) | 65 | 42 | 37 | 2 | 32 | 16
Neutrophil count decreased (Investigations) | 64 | 21 | 20 | 2 | 15 | 9
Platelet count decreased (Investigations) | 23 | 5 | 1 | 0 | 8 | 2
Weight decreased (Investigations) | 25 | 1 | 3 | 0 | 1 | 2
White blood cell count decreased (Investigations) | 22 | 11 | 5 | 0 | 7 | 5
Decreased appetite (Metabolism and nutrition disorders) | 17 | 3 | 4 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4 | 3 | 1 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 5 | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1 | 4 | 0 | 1 | 3
Headache (Nervous system disorders) | 27 | 6 | 10 | 2 | 3 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 3 | 2 | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 2
Seizure (Nervous system disorders) | 5 | 0 | 0 | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 13 | 5 | 1 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 5 | 2 | 0 | 0 | 0 | 2
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 1 | 0 | 1 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 5 | 5 | 1 | 0 | 1 | 3
Vulvovaginal pruritus (Reproductive system and breast disorders) | 5 | 4 | 2 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 50 | 7 | 14 | 2 | 9 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 2 | 4 | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 4 | 1 | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1 | 0 | 2 | 2
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 17 | 1 | 2 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 18 | 4 | 8 | 0 | 5 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 9 | 1 | 1 | 0 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 9 | 3 | 1 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 3 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 11 | 1 | 2 | 1 | 1 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 8 | 2 | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No